CLINICAL TRIAL: NCT02275416
Title: Safety of UV1 Vaccination in Combination With Ipilimumab in Patients With Unresectable or Metastatic Malignant Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ultimovacs ASA (Industry)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UV1/hTERT-MM; 2013-005582-39 (EudraCT Number)
Record Dates: First submitted 2014-09-12; First posted 2014-10-27 (Estimated); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; UV1 vaccine; Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ipilimumab & UV1 vaccine & GM-CSF (Experimental): Ipilimumab (3 mg/kg) every 3rd week for a total of 4 doses. GM-CSF (75 μg) followed by UV1 vaccine (300 μg) will be injected intradermally in the lower abdomen before and between treatments of ipilimumab and thereafter every 4th week up to 28 weeks, and thereafter at week 36 and 48.
  Interventions: Drug: Ipilimumab; Biological: UV1 vaccine; Biological: GM-CSF

INTERVENTIONS:
Drug: Ipilimumab
  Other Names: Yervoy
Biological: UV1 vaccine
  Other Names: UV1
Biological: GM-CSF
  Other Names: Leukine

SUMMARY:
This study, with 20 patients participating, will examine the safety and tolerability for the ipilimumab/UV1 combination in patients with unresectable or metastatic malignant melanoma.

DETAILED DESCRIPTION:
This is a phase I/IIa, national, open label, single arm, interventional study examining safety and tolerability for the ipilimumab/UV1 combination in patients with unresectable or metastatic malignant melanoma. Patients that have signed the informed consent form will be asked to take part in the study. All patients will receive ipilimumab together with the UV1 vaccine and rranulocyte-macrophage colony-stimulating factor (GM-CSF). Ipilimumab will be given every 3rd week for a total of 4 doses. The UV1 vaccine and GM-CSF will be given before and between treatments of ipilimumab. The maximum number of UV1/GM-CSF will be 10 doses.

Immunoresponders maybe followed up every third months for 5 years after the first UV1 treatment. Follow-up is onging.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of unresectable or metastatic malignant melanoma, including cutaneous, ocular, mucosal and unknown primary tumour.
2. Unresectable Stage III or Stage IV melanoma (AJCC 2010)
3. Prior adjuvant melanoma therapy is permitted; any number of previous treatments for melanoma is permitted.
4. ECOG performance status of 0 or 1 (see Error! Reference source not found.).
5. Men and women ≥ 18 years of age
6. Adequate hematologic, renal and hepatic function, specifically:

   1. WBC ≥ 2500/μL
   2. Absolute neutrophil count (ANC) ≥ 1000/uL
   3. Platelets ≥ 75 x 103/μL
   4. Haemoglobin ≥ 9 g/dL
   5. Creatinine ≤ 2.5 x ULN
   6. AST/ALT ≤ 3 x ULN for patients without liver metastasis; ≤ 5 x ULN for patients with liver metastasis
   7. Total bilirubin ≤ 3 x ULN, (except patients with Gilbert's Syndrome, who must have a total bilirubin less than 3.0 mg/dL)
7. Women of childbearing potential and men must be using an acceptable method as described in the protocol to prevent pregnancy.
8. Signed informed consent and expected cooperation of the patients for the treatment and follow up must be obtained and documented according to ICH GCP, and national/local regulations.

Exclusion Criteria:

1. History of or current active autoimmune diseases, including but not limited to inflammatory bowel diseases, rheumatoid arthritis, autoimmune thyroiditis, autoimmune hepatitis, systemic sclerosis (scleroderma and variants), systemic lupus erythematosus, autoimmune vasculitis, autoimmune neuropathies (e.g. Guillain-Barre syndrome). Patients with vitiligo are not excluded.
2. MRI detected active brain metastasis witch require other therapies such as surgery and/or radiation therapy. Patients already treated for their brain metastasis, surgery or radiation therapy, and have had stable disease for more than two month and NOT requiring steroids may however be included in this study.
3. Uncontrolled infectious diseases - requires negative tests for clinically suspected human immunodeficiency virus (HIV), hepatitis B virus (HBV) and hepatitis C virus (HCV).
4. History of or current immunodeficiency disease, splenectomy or splenic irradiation
5. Prior allogeneic stem cell transplantation
6. Pregnancy
7. Women who are breastfeeding
8. Any underlying medical or psychiatric condition, which in the opinion of the Investigator, will make the administration of study drug hazardous or obscure the interpretation of Adverse Events, such as a condition associated with frequent diarrhoea
9. History of allergic reaction to parenteral administered recombinant protein product
10. History of another malignancy that in the opinion of the investigator may compromise the outcome of the study
11. Any reason why, in the opinion of the investigator, the patient should not participate.
12. Known serious reactions or hypersensitivity to any components of the UV1 vaccine or similar peptide based vaccines
13. Known hypersensitivity to GM-CSF
14. Known hypersensitivity to any of the excipients of the investigational products
15. Concomitant use of antithrombotic agents with the exception of platelet inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-02-02 (Actual); Primary Completion 2016-10-06 (Actual); Study Completion 2020-11-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability profile. Frequency/ severity of adverse and serious adverse events. Biochemistry and hematology results, vital signs and ECOG | Up to 53 weeks
  Frequency and severity of adverse events and serious adverse events. Biochemistry and hematology results, vital signs and ECOG performance status will be assessed.

SECONDARY OUTCOMES:
Immunological response. Number of T-cell responses including time to T-cell response, level of response and duration of response. | Up to 53 weeks
  Number of T-cell responses including time to T-cell response, level of response and duration of response.
Treatment response. Tumour response evaluated by CT scan every 12th week. | Up to 48 weeks
  Tumour response evaluated by CT scan every 12th week.
Health Related Quality of Life (HRQL) | Up to 53 weeks
  HRQL measured by use of patient questionnaire EORTC QLQ-C30

OTHER OUTCOMES:
Explore potential biomarkers for efficacy and safety of the ipilimumab/UV1 combination | Up to 48 weeks
  Exploratory biomarker analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Tormod Guren, MD PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Radiumhospitalet, Oslo, Norway

REFERENCES:
- [Derived] Ellingsen EB, Bounova G, Kerzeli I, Anzar I, Simnica D, Aamdal E, Guren T, Clancy T, Mezheyeuski A, Inderberg EM, Mangsbo SM, Binder M, Hovig E, Gaudernack G. Characterization of the T cell receptor repertoire and melanoma tumor microenvironment upon combined treatment with ipilimumab and hTERT vaccination. J Transl Med. 2022 Sep 11;20(1):419. doi: 10.1186/s12967-022-03624-z. PMID 36089578
- [Derived] Aamdal E, Inderberg EM, Ellingsen EB, Rasch W, Brunsvig PF, Aamdal S, Heintz KM, Vodak D, Nakken S, Hovig E, Nyakas M, Guren TK, Gaudernack G. Combining a Universal Telomerase Based Cancer Vaccine With Ipilimumab in Patients With Metastatic Melanoma - Five-Year Follow Up of a Phase I/IIa Trial. Front Immunol. 2021 May 11;12:663865. doi: 10.3389/fimmu.2021.663865. eCollection 2021. PMID 34046035